CLINICAL TRIAL: NCT02269826
Title: Medical Device Study to Investigate the Efficacy and Tolerability of Vagisan® Moisturising Cream vs. Gynomunal® Vaginal Gel in a 2-period Changeover Design in n=120 Patients With Vaginal Dryness Who Cannot or do Not Wish to Use Oestrogens
Brief Title: Efficacy and Safety of Non-hormonal Vaginal Preparations in Treating Vaginal Dryness
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dr. August Wolff GmbH & Co. KG Arzneimittel (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: LB-04/2007
Record Dates: First submitted 2014-10-14; First posted 2014-10-21 (Estimated); Last update posted 2018-02-19 (Actual); Status verified 2018-02

CONDITIONS: Vaginal Dryness

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Vagisan® Moisturising Cream (Experimental): non-hormonal vaginal cream for the treatment of vulvovaginal dryness
  Interventions: Device: Vagisan® Moisturising Cream
- Gynomunal® vaginal gel (Active Comparator): non-hormonal gel
  Interventions: Device: Gynomunal® vaginal gel

INTERVENTIONS:
Device: Vagisan® Moisturising Cream — Once in the evenings before going to bed, intravaginally with the help of the applicator included (approximately 2.5 g per application) and perivaginally one fingertip unit (approximately 0.5 g per application).
  Other Names: WO 2085
  Arms: Vagisan® Moisturising Cream
Device: Gynomunal® vaginal gel — Once in the evenings before going to bed, intravaginally with the help of the applicator included (approximately 2.5 g per application) and perivaginally one fingertip unit (approximately 0.5 g per application).
  Arms: Gynomunal® vaginal gel

SUMMARY:
Vulvovaginal irritation due to dryness is a frequent complaint among post- and some premenopausal women. International guidelines recommend non-hormonal products as first line therapy.

Efficacy and safety of the medical device Vagisan® Moisturising Cream (VMC), a non-hormonal vaginal cream for the treatment of vulvovaginal dryness and Gynomunal Vaginal Gel (GVG), a non-hormonal gel should be compared in a 12-week multicentre, open-label, randomised, two-period cross-over phase III trial. The hypothesis was that VMC is non-inferior to GVG.

The primary endpoint was the sum of subjective symptoms of vulvovaginal atrophy (VVA) added up over each treatment period. Furthermore, objective symptoms of VVA and adverse effects were planned to be assessed. 120 women should be randomly allocated to either of the two treatments, each given over a period of 4 weeks.

DETAILED DESCRIPTION:
The purpose of the study was to test the non-inferiority of the medical device Vagisan® Moisturising Cream (VMC) in comparison to Gynomunal® vaginal gel (GVG) in 6 centres in 120 women who suffered from "vaginal dryness". The main objective criterion was to compare the sum of 4 subjective symptoms of "vaginal dryness" measured daily over a period of 28 days. VMC should be applied daily, while GVG had to be administered daily during the first week and twice weekly thereafter.

The main objective parameter for efficacy analysis was the sum of the subjective symptoms of vaginal dryness (feeling of dryness, itching, burning sensation and pain) before, during (patient diaries) and after the 28-day therapy period.

The per-protocol analysis and of the intent-to-treat analysis should prove non-inferiority of VMC compared to GVG, despite a possible carry-over effect to the detriment of VMC. To avoid the problem of any possible carry-over effect the analysis of the first period was chosen for the primary comparison of both products.

Furthermore, objective symptoms of vaginal dryness detected via colposcopy, the vaginal secretion's pH, the efficacy assessment by the patients and the treating doctor and patients' questionnaires with regard to the product characteristics of the medical devices should be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Women over the age of 18.
* Women with vaginal dryness who do not want to or are not allowed to use oestrogens, such as post-menopausal women, women with oestrogen-dependent tumours in their medical history and women who had been treated with systemic medicinal products that can have a drying-out effect on the vaginal mucous membranes.
* Total score (0-16) of at least 3 of four subjective symptoms (feeling of dryness, itching, burning sensation and pain).
* Written declaration of consent for the voluntary participation in the study is present.

Exclusion Criteria:

* Known hypersensitivity to one of the ingredients of the test and/or reference medical device.
* Current vaginal infections.
* Recurring (i.e. at least 3) vaginal infections within the last 12 months.
* Additional (not study-related) treatment of vaginal dryness during the therapy phases.
* Therapy with antibiotics, steroids (excluding sexual steroids in oral, dermal or transdermal application) or antimycotics in the last 14 days before inclusion and participation in this study.
* Women who are not able to participate properly in this study.
* Fertile women without sufficient contraceptive protection.
* Fertile women who are pregnant (positive HCG test) or breastfeeding.
* Current alcohol and/or drug abuse.
* Participation in another clinical study within the last four weeks and/or parallel participation in this study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 117 (Actual)
Dates: Start 2008-02; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
per patient intraindividually determined total score consisting of the patients' subjective symptoms (feeling of dryness, itching, burning sensation and pain) | Therapy period of 28 days
  The main objective criterion for the confirmatory analysis was the per patient intraindividually determined total score consisting of the patients' subjective symptoms (feeling of dryness, itching, burning sensation and pain, each rated as 0=not present, 1=hardly pronounced, 2=moderately pronounced, 3=quite pronounced, 4=very pronounced) during the course of therapy. This was based on the daily entry in the patient diary.

SECONDARY OUTCOMES:
Intraindividually determined total score consisting of the evaluations of the objective "vaginal dryness" diagnoses | 28 days
  • Descriptive account of the per patient intraindividually determined total score consisting of the evaluations of the objective "vaginal dryness" diagnoses made by the investigator during the visits (thinning of the epithelium, redness, petechial bleeding, discharge, each rated as 0=not present, 1=hardly pronounced, 2=moderately pronounced, 3=quite pronounced, 4=very pronounced).
Patients' individual subjective symptoms of "vaginal dryness" | 28 days
  Descriptive account of the patients' individual subjective symptoms of "vaginal dryness" expressed during the visits (feeling of dryness, itching, burning sensation and pain).
Overall efficacy and tolerability assessments | 28 days
  The overall efficacy and tolerability assessments (investigator and/or patient) with the ratings "very good", "good", "satisfactory" and "poor".
Occurrence of side effects | 28 days
  The assessment of one-sided 95% confidence intervals for the occurrence of side effects when using the test and reference medical device
Assessment of adverse events | 28 days
  The assessment of adverse events that have not been classified as related to the medical device.
Vaginal pH | 28 days
  Descriptive account of the vaginal pH as determined by the investigator during the visits.
Patients' subjective satisfaction with the test and reference medical device | 28 days
  The patients' subjective satisfaction with the test and reference medical device based on a patient questionnaire conducted at the end of each treatment period [feeling of skin (within approximately 10 minutes of application and the following morning), discharge the next morning, stickiness, spreadability on the vulva (perivaginal), cooling effect, softness of the medical device, fragrance, handling of the applicator, overall assessment by the sexual partner] with ratings from 1 (very positive) to 6 (very negative) or 0=no assessment (see chapter 9.1.6 "Patient questionnaire").

CONTACTS AND LOCATIONS:
Overall Officials: Christoph Abels, Prof., MD, Study Director — Dr. August Wolff GmbH & Co. KG Arzneimittel; Klaus-Michael Grunwald, MD, Principal Investigator
Locations (6):
- Germany (6):
  - Dr. med. Kirsten Grunwald, Aachen
  - Dr. med. Julia Wanke, Aachen
  - Dr. med. Axel Gerick, Aachen
  - Dr. med. Ralf Conrads, Aachen
  - Wolfgang Clemens, Stolberg
  - Anja Obermeyer, Würselen

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Stute P, May TW, Masur C, Schmidts-Winkler IM. Efficacy and safety of non-hormonal remedies for vaginal dryness: open, prospective, randomized trial. Climacteric. 2015;18(4):582-9. doi: 10.3109/13697137.2015.1036854. Epub 2015 May 22. PMID 25845406